CLINICAL TRIAL: NCT02778035
Title: A Randomized Controlled Trial Comparing Different Patterns of Repetitive Transcranial Magnetic Stimulation in the Treatment of Refractory Depression
Brief Title: Comparing Different Patterns of rTMS in Major Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-9615
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: Depression; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- 60 min inter-session interval (Experimental): Repetitive transcranial magnetic stimulation (rTMS) to bilateral dorsomedial prefrontal cortex, twice daily, 5 days per week for 4 weeks (Inter-session interval, 60 min).
  Interventions: Device: Dorsomedial prefrontal rTMS
- 30 min inter-session interval (Experimental): Repetitive transcranial magnetic stimulation (rTMS) to bilateral dorsomedial prefrontal cortex, twice daily, 5 days per week for 4 weeks (Inter-session interval, 30 min).
  Interventions: Device: Dorsomedial prefrontal rTMS
- 0 min inter-session interval (Experimental): Repetitive transcranial magnetic stimulation (rTMS) to bilateral dorsomedial prefrontal cortex, twice daily, 5 days per week for 4 weeks (Inter-session interval, 0 min).
  Interventions: Device: Dorsomedial prefrontal rTMS

INTERVENTIONS:
Device: Dorsomedial prefrontal rTMS — Dorsomedial prefrontal rTMS, bilateral, iTBS, 600 pulses per hemisphere, 120% RMT, 2 sessions at 0, 30, or 60 min inter-session interval

SUMMARY:
This trial will compare the trajectories of improvement for three different patterns of twice-daily rTMS in major depression: two daily sessions of dorsomedial prefrontal rTMS delivered at 0 min vs. 30 min vs. 60 min intervals.

ELIGIBILITY:
Participants are eligible for the study if they:

1. are outpatients
2. are voluntary and competent to consent to treatment
3. have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of major depressive disorder (MDD), single or recurrent, or Bipolar Disorder with a current Major Depressive Episode
4. are between the ages of 18 and 65
5. have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of > 3 in the current episode OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF 1 or 2)
6. have a score ≥18 on the 17-item Hamilton Rating Scale for Depression (HRSD-17)
7. have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
8. are able to adhere to the treatment schedule
9. pass the TMS safety-screening questionnaire
10. have normal thyroid functioning and no clinically significant abnormalities on complete blood count (CBC), on pre-study blood work.

Participants are ineligible for the study if they:

1. have a history of substance dependence or abuse within the last 3 months
2. have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
3. have active suicidal intent
4. are pregnant
5. have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
6. have a MINI diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, assessed by a study investigator to be primary and causing greater impairment than MDD
7. have a diagnosis of any personality disorder, and assessed by a study investigator to be primary and causing greater impairment than MDD
8. have failed a course of electroconvulsive therapy (ECT) in the current episode or previous episode
9. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
10. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
11. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
12. have a clinically significant laboratory abnormality, in the opinion of the investigator
13. currently (or in the last 4 weeks prior to the study) have taken more than lorazepam 4 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
14. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
17-Item Hamilton Rating Scale for Depression (HAMD-17) | Baseline, after each week of treatment (i.e. after 5 days of treatment), and 1, 4, and 12 weeks post-treatment. Treatment will include 5 daily weekday visits over 4 weeks (20 sessions total).
  Outcome measured by a change in HAMD-17 score from baseline to 1-week post-treatment. A 50% improvement in the score is considered a response to rTMS. A final score of ≤7 is categorized as remission.

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | Daily for 4 weeks, 5 days per week, in addition to three follow-up visits at 1, 4, and 12 weeks post-treatment
  Outcome measured by a change in BDI-II score from baseline to 1-week post-treatment. A 50% improvement in the score is considered a response to rTMS. A final score of ≤12 is categorized as remission.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - UHN MRI-Guided rTMS Clinic, Toronto Western Hospital, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- [Derived] Goodman MS, Schulze L, Daskalakis ZJ, Konstantinou GN, Mansouri F, Trevizol AP, Blumberger DM, Downar J. Randomised controlled trial comparing different intersession intervals of intermittent theta burst delivered to the dorsal medial prefrontal cortex. BMJ Ment Health. 2024 Oct 23;27(1):e301290. doi: 10.1136/bmjment-2024-301290. PMID 39448077